CLINICAL TRIAL: NCT02758964
Title: Evaluation of Cerebral Thrombembolism After TAVR
Acronym: EARTH - TAVR
Status: Completed | Type: Observational
Sponsor: Charite University, Berlin, Germany (Other)
Collaborators: Bayer (Industry)
Responsible Party: Principal Investigator, Ulf Landmesser, Prof. Dr. Ulf Landmesser, Charite University, Berlin, Germany
Other Study IDs: EARTH - TAVR 01
Record Dates: First submitted 2016-04-24; First posted 2016-05-03 (Estimated); Last update posted 2019-04-02 (Actual); Status verified 2019-03

CONDITIONS: Aortic Valve Stenosis; Transcatheter Aortic Valve Replacement; Intracranial Embolism
Keywords: TAVR; TAVI; Transcatheter Aortic Valve Replacement; Intracranial Embolism
MeSH Terms: conditions — Aortic Valve Stenosis; Intracranial Embolism | interventions — Magnetic Resonance Spectroscopy

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes

INTERVENTIONS:
Other: MRI, neurocognitive Testing — A cerebral MRI and neurocognitive testing will be performed before TAVR, before hospital discharge and after 3 months

SUMMARY:
EARTH-TAVR is a diagnostic multicenter study to evaluate the occurrence and extent of cerebral embolization (total new lesion volume) in patients before TAVR versus 3 months after TAVR.

DETAILED DESCRIPTION:
Calcific aortic valve stenosis is the most common cause of aortic stenosis (AS) among adults in Europe and in the United States. The prevalence of moderate or severe AS was found to be age-dependent rising from 0.02% in patients aged 18-44 years to 2.8% in patients aged ≥ 75 years. Among patients at prohibitive surgical risk, TAVR has become the treatment of choice.The safety and efficacy of TAVR compared with medical management and SAVR has been demonstrated in clinical trials.The composite of the rate of all-cause death or stroke was 27% and 37% in TAVR patients after 1 and 2 years, respectively.Even though parts of the strokes occur during the peri-procedural period, the patients remain at risk of stroke throughout the first months after the procedure.

EARTH-TAVR is a diagnostic multicenter study performing in association with the GALILEO trial (NCT02556203), which is investigating cerebral embolization with MRI and neurocognitive testing in patients undergoing TAVR, who are treated with anticoagulation (Rivaroxaban/ASS) or DAPT (Clopidogrel/ASS). GALILEO is a global multicenter, open-label, randomized, event-driven, active-controlled study comparing a rivaroxaban-based antithrombotic strategy to an antiplatelet-based strategy after transcatheter aortic valve replacement (TAVR) to optimize clinical outcomes.

Investigators aim to investigate peri-interventional and delayed cerebral embolization in the early period (3 months) after TAVR and to analyze associations between neurocognitive parameters and cerebral embolization patterns in patients on different antithrombotic treatment regimes.

ELIGIBILITY:
Inclusion Criteria:

* Man or woman of 18 years of age or older
* Via iliofemoral or subclavian access
* Provide written IC

Exclusion Criteria:

* Atrial fibrillation (AF), current or previous, with an ongoing indication for oral anticoagulant Treatment
* Any other indication for continued treatment with any oral anticoagulant (OAC)
* Known bleeding diathesis (such as but not limited to active internal bleeding, clinically significant bleeding, platelet count ≤ 50,000/mm3 at screening, hemoglobin level < 8.5 g/dL, active peptic ulcer or known gastrointestinal (GI) bleeding, history of intracranial hemorrhage or subdural hematoma)
* Any indication for dual-antiplatelet therapy (DAPT) for more than 3 months after randomization (such as coronary, carotid or peripheral stent implantation)
* Clinically overt stroke within the last 3 months
* Planned coronary or vascular intervention or major surgery
* Severe renal impairment (eGFR < 30 mL/min/1.73 m2) or on dialysis, or post-TAVR unresolved acute kidney injury with renal dysfunction stage 2 or higher
* Moderate and severe hepatic impairment (Child-Pugh Class B or C) or any hepatic disease associated with coagulopathy
* Any contraindication for cerebral MRI, in particular:
* non-MRI-conditional pacemakers
* MRI conditional pacemakers <4 weeks after implant
* any metal fragments in the eye
* aneurysm clip in the brain
* severe claustrophobia

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients 18 years or older wirth aortic valve stenosis receiving TAVR-Intervention.
Sampling Method: Probability Sample
Enrollment: 55 (Actual)
Dates: Start 2016-09; Primary Completion 2019-01 (Actual); Study Completion 2019-01 (Actual)

PRIMARY OUTCOMES:
Total volume of new cerebral lesions on MRI, 3 months after TAVR versus Baseline | 3 months after TAVR versus baseline
  Occurrence and extent of cerebral embolization in patients after TAVR measured by total volume of new ischemic cerebral lesions on DWI and FLAIR MRI.
  Total new lesion volume is defined as the sum volume of all new cerebral ischemic lesions on the 3 months post-procedural MRI relative to the pre-TAVR cerebral MRI scan (on diffusion weighted and FLAIR MRI images)

SECONDARY OUTCOMES:
New lesion volume of cerebral embolization in patients treated with ASS and rivaroxaban 10mg OD versus an antiplatelet -based strategy with ASS and clopidogrel. | 3 months post TAVR versus baseline
  Total new lesion volume is defined as the sum volume of all new cerebral ischemic lesions on the 3 months post-procedural MRI relative to the pre-TAVR cerebral MRI scan (on diffusion weighted and FLAIR MRI images).
extent and location of new cerebral lesions early AFTER TAVR and after 3 months | MRI after TAVR (0-7 days after TAVR) compared to 3 months after TAVR
  To evaluate cerebral embolisation, which is not procedure related, cerebral embolisation on MRI will be compared 3 months post TAVR versus the post-TAVR MRI scan
Assessment of different neurocognitive tests (NIHSS-score, MOCA-score, MOT-score, PAL-score, RTI-score, SWM-score, AST-score, CAM-Score); change of sum scores before, after and 3 months after TAVR procedure. | Before TAVR, post TAVR and after 3 months
  To evaluate neurologic function with a battery of neurocognitive tests and to correlate these findings to cerebral MRI scans
Extent and localization of clinically apparent non-cerebral emboli after TAVR | baseline, post TAVR and after 3 months
  To describe extent and localization of non-cerebral embolisation (e.g. pulmonary embolism, limb ischaemia...)
Evaluation of possible changes in quality of life after TAVI with EQ-5D questionnaire sum score. | Baseline versus 3 months following TAVR

CONTACTS AND LOCATIONS:
Overall Officials: Ulf Landmesser, Prof. Dr., Principal Investigator — Charité - Universitätsmedizin Berlin, Department of Cardiology; Matthias Endres, Prof. Dr., Study Chair — Charité - Universitätsmedizin Berlin, Department of Neurology; Georg M Fröhlich, PD, Study Chair — Charité - Universitätsmedizin Berlin, Department of Cardiology; Volkmar Falk, Professor, Study Chair — German Heart Institute
Locations (2):
- Germany (2):
  - Charité - Universitätsmedizin Berlin, Campus Mitte, Berlin
  - Charité - Universitätsmedizin Berlin, Campus Benjamin Franklin, Berlin

REFERENCES:
- [Background] Holmes DR Jr, Brennan JM, Rumsfeld JS, Dai D, O'Brien SM, Vemulapalli S, Edwards FH, Carroll J, Shahian D, Grover F, Tuzcu EM, Peterson ED, Brindis RG, Mack MJ; STS/ACC TVT Registry. Clinical outcomes at 1 year following transcatheter aortic valve replacement. JAMA. 2015 Mar 10;313(10):1019-28. doi: 10.1001/jama.2015.1474. PMID 25756438
- [Background] Osnabrugge RL, Mylotte D, Head SJ, Van Mieghem NM, Nkomo VT, LeReun CM, Bogers AJ, Piazza N, Kappetein AP. Aortic stenosis in the elderly: disease prevalence and number of candidates for transcatheter aortic valve replacement: a meta-analysis and modeling study. J Am Coll Cardiol. 2013 Sep 10;62(11):1002-12. doi: 10.1016/j.jacc.2013.05.015. Epub 2013 May 30. PMID 23727214
- See also: GALILEO main study — http://www.cardialysis.com/galileo/
- See also: GALILEO study — https://clinicaltrials.gov/ct2/show/NCT02556203?term=GALILEO&rank=7